CLINICAL TRIAL: NCT05417542
Title: Multimodal Analysis of the Young Brain on Rhythm Perception: From Premature Neonates to Infants
Acronym: Exposition
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PI2021_843_0054
Record Dates: First submitted 2022-05-31; First posted 2022-06-14 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Time Perception; Rhythm; EEG; fNIRS; ERP; Premature Neonates; Discrimination
Keywords: Time perception; rhythm; EEG; fNIRS; ERP; Premature neonates; Discrimination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Exposition I (Experimental): preterm neonates between 28 and 30 wGA Exposition to music during the NICU period
  Interventions: Other: EEG; Other: NIRS
- Exposition II (Experimental): preterm neonates between 32 and 34 wGA Exposition to music during the NICU period
  Interventions: Other: EEG; Other: NIRS
- Control I (Active Comparator): preterm neonates between 28 and 30 wGA
  Interventions: Other: EEG; Other: NIRS
- Control II (Active Comparator): preterm neonates between 32 and 34 wGA
  Interventions: Other: EEG; Other: NIRS
- Control III (Active Comparator): preterm neonates between 36 and 40 wGA
  Interventions: Other: EEG; Other: NIRS

INTERVENTIONS:
Other: EEG — EEG recording during prematurity or around term
Other: NIRS — NIRS recording during prematurity or around term

SUMMARY:
Premature neonates are able to discriminate phonemes and voice from 28wGA at a time the neuronal network establish contact between the environment and the cortical neurones. In the present monocentric study the investigators will analyse the response of the cortical network in premature aged between 28 and 40 wGA in response to auditory stimuli using High Resolution Electroencephalography and High Density Near Infrared Spectroscopy

ELIGIBILITY:
Inclusion Criteria:

* Full term neonates between 28 and 40 weeks Gestational Age

Exclusion Criteria:

* Neonates outside the age range

Ages: 0 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-05-31 (Actual); Primary Completion 2029-05 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Variations of the response of the cortical network using High Resolution Electroencephalography before auditory stimuli between the 5 infant groups | one day
Variations of the response of the cortical network using High Resolution Electroencephalography during auditory stimuli between the 5 infant groups | one day
Variations of the response of the cortical network using High Resolution Electroencephalography after auditory stimuli between the 5 infant groups | one day
variations of the response of the cortical network using High Density Near Infrared Spectroscopy before auditory stimuli between the 5 infant groups | one day
variations of the response of the cortical network using High Density Near Infrared Spectroscopy during auditory stimuli between the 5 infant groups | one day
variations of the response of the cortical network using High Density Near Infrared Spectroscopy after auditory stimuli between the 5 infant groups | one day

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No